CLINICAL TRIAL: NCT06704880
Title: Lower Limb Constraint-induced Movement Training Versus Strength Training of the Non-hemiplegic Lower Limb on Motor Performance in Children With Hemiplegic Cerebral Palsy: A Randomized Control Trial.
Brief Title: CONSTRAINT-INDUCED MOVEMENT THERAPY VERSUS CROSS EDUCATION IN CHILDREN WITH CEREBRAL PALSY
Acronym: NEUROLOGY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Abdullah Owaid Kerdi Alanazi, PHYSIOTHERAPIST, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-PGS-2024-03-156
Record Dates: First submitted 2024-09-09; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hemiplegic Cerebral Palsy
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIMT GROUP (Experimental)
  Interventions: Other: rehabilitation
- STRENGHTH TRAINING GROUP (cross education) (Experimental)
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — children in the CIMT group will RECIEVE lower limb CIMT for the non-hemiplegic limb using whole leg orthosis. Children in cross-education group will receive strengthening training for the non-hemiplegic lower limb

SUMMARY:
This clinical trial aims to Compare the effectiveness of lower limb CIMT and the Strength Training of the Non-Hemiplegic lower limb on motor performance in hemiplegic children with CP.

Participants will:

diagnosed with hemiplegic cerebral palsy treated with CIMT or Strength training (cross-education) for a non-hemiplegic limb for 8 weeks.

3 sessions per week. Measurements will be taken at baseline and then at the end of the 8 weeks.

DETAILED DESCRIPTION:
Method:

32 children with hemiplegic CP will be equally and randomly allocated to two groups (group A and B). group A will receive lower limb CIMT for the non- hemiplegic limb using whole leg orthosis and Group B will receive strengthen training for the non-hemiplegic lower limb. Both groups will receive routine physical therapy for the hemiplegic lower limb. Both groups will receive 60 minutes training session for 3 sessions per week for 8 consecutive weeks. Assessment will be at baseline then at the end of trial.

ELIGIBILITY:
Inclusion Criteria:

1. Children with hemiplegic cerebral palsy aged age between 4 and 10.
2. (GMFCS) levels I, II and III.
3. Able to follow therapist instructions during training session.

Exclusion Criteria:

1. Lack of patient's cooperation.
2. Difficulty wearing constraint method due to severe joint deformation or/and contracture.
3. Patients were treated with botulinum toxin during the last 3 months.
4. Seizure disorder not fully controlled by medication.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
gait speed | at base line then at the end of the 8 weeks
  gait spatiotemporal parameter
cadence gait spatiotemporal parameter | at base line then at the end of the 8 weeks
  gait spatiotemporal parameter
step length | at base line then at the end of the 8 weeks
  gait spatiotemporal parameter
stride length | at base line then at the end of the 8 weeks
  gait spatiotemporal parameter

SECONDARY OUTCOMES:
Pediatric balance scale | at base line then at the end of the 8 weeks
  Pediatric balance scale The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
6 Minute walk test (6MWT) | at base line then at the end of the 8 weeks
  endurance measurement
Modified Ashworth scale | at base line then at the end of the 8 weeks
  measuring muscle tone Scoring 0 No Increased in tone
  1. Slight increase in tone giving a catch when the limb is moved in flexion or extension 1+ Slight increase in muscle tone, indicated by a catch followed by minimal resistance throughout range of motion (ROM)
  2. More marked increase in tone through most of the ROM, but the limb easily flexed
  3. Considerable increase in tone, passive movement difficult
  4. Limb rigid in flexion or extension
Handheld dynamometer | at base line then at the end of the 8 weeks
  measuring muscles strength

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahmn Alfaisal University, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No